CLINICAL TRIAL: NCT06218576
Title: Sensitivity Comparison of Follow-up MRI Between Acute Cerebral and Cerebellar Cortical Microinfarctions ( CMI )
Brief Title: Sensitivity Comparison of Follow-up MRI Between Acute Cerebral and Cerebellar Cortical Microinfarctions ( CMI )Microinfarctions
Acronym: CMI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2023/DR-01
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Acute Cerebral and Cerebellar Cortical Microinfarctions (CMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute cerebral and/or cerebellar CMI: Patients with acute cerebral and/or cerebellar CMI
  Interventions: Other: None, purely observational study

INTERVENTIONS:
Other: None, purely observational study — None, purely observational study

SUMMARY:
Cerebral cortical microinfarctions (CMI) are frequently observed on MRI and histology studies, especially in elderly patients and in patients with cognitive dysfunction. The majority of these studies analysed chronic cerebral CMI lesions.

The few studies reporting on temporal dynamics of MRI signal of acute cerebral CMI showed very low sensibility for persisting signal changes on follow-up MRI on standard MRI sequences. A retrospective study, analysing follow-up 3T MRI in 25 patients with acute cerebral CMI (defined as ≤10 mm on DWI), showed a chronic cerebral CMI detection rate of only 16% on T2-weighted and 5% on FLAIR imaging after a mean follow-up period of 33 months (with a very wide range of 0.5-142 months). Another 3T MRI study including seven patients showed disappearance of all acute cerebral very small-sized CMI (defined as <5 mm size on initial DWI) on all follow-up MRI sequences (T1- and T2-weighted and FLAIR imaging, performed after one month).

Recently, it has been shown that chronic relatively small (<20 mm) cerebellar cortical infarctions (based on diffusion-weighted imaging) were frequently observed in acute stroke patients, especially in case of cardioembolic stroke (with chronic small cerebellar cortical infarctions observed in 32% of cases). The high prevalence of these chronic small cerebellar cortical infarctions suggest a possible higher detection rate of chronic small-sized infarction in the cerebellum compared to the supratentorial brain.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to our stroke centre between February 2021 and June 2023 with the following inclusion criteria:

* age >18 years,
* initial MRI performed within one week after symptom onset,
* symptomatic brain infarction confirmed by DWI,
* presence of acute cerebral and/or cerebellar CMI

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient admitted to Nîmes University Hospital between February 2021 and June 2023 with initial MRI performed within one week after symptom onset, symptomatic brain infarction confirmed by DWI, and the presence of acute cerebral and/or cerebellar CMI
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Chronic CMI | 6 monthes
  Detection rate of chronic CMI on follow-up MRI used in daily clinical practice after initial acute cerebral and cerebellar CMI (≤10 mm) (Nb)
CMI localisations | 6 monthes
  Compare initial acute cerebral and cerebellar CMI (≤10 mm) localisation (cerebral or cerebellar)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France